CLINICAL TRIAL: NCT04217824
Title: a Prospective, Randomized, Double-blind Study. comparıson of Karydakis Flap and Limberg Flap Treatment of Pilonidal Sinus in Adolescent. a Prospective, Randomised Study
Brief Title: Comparison of Karydakis and Limberg Flap Treatment of Pilonidal Sinus in Adolescent. a Prospective, Randomised Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Ahmet Gökhan Güler, assistant professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2019/04-02
Record Dates: First submitted 2020-01-02; First posted 2020-01-03 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Pilonidal Sinus; Postoperative Complications
Keywords: pilonidal sinus; presakral apse; limberg flap; karydakis flap
MeSH Terms: conditions — Pilonidal Sinus; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- karydakis flap (Active Comparator): An asymmetric elliptical excision is performed, defective tissues between the lower and upper ends are removed until they reach healthy borders. The wound edge is then mobilized and the flap is slid over the corresponding wound edge by suturing to the fascia and the skin to the appropriate wound layers. Thus, the gluteal groove is lateralized. Subcutaneous tissue and skin are closed.
  Interventions: Procedure: pilonidal sinus excision
- limberg flap (Active Comparator): Rhomboid excision and pilonidal sinuses together with damaged tissue. On the right side of the patient, the intact skin is shifted to the medial area where the tissues are removed without tension. Thus, the defective part and gluteal groove are corrected.
  Interventions: Procedure: pilonidal sinus excision

INTERVENTIONS:
Procedure: pilonidal sinus excision — Closure of the defect in pilonidal sinus excision with one of the randomly selected flap methods.

SUMMARY:
Pilonidal sinus disease (PSD) is a chronic inflammation and infection of the sacrococcygeal region. Produces clinic findings with abscess and discharge in the sacrococcygeal region or painful sinus tract in the natal cleft. Its incidence rate among Turkish servicemen is reported to be 8.8% in a study. Although pilonidal sinus disease is common in men, this is the opposite in adolescence. Because adolescent girls are 2 or 3 times more.

Karydakis flap and Limberg flap operations widely preferred in recent years in the surgical treatment of PSD. In our study, we aim to compare these two techniques prospectively and randomly.

DETAILED DESCRIPTION:
The best treatment technique for pilonidal sinus disease (PSD) is still controversial. While some researchers prefer minimally invasive methods, some researchers prefer surgical treatment. The most important concern in surgical treatment options is the prolongation of the disease recovery time and recurrence of the disease. Complications that may develop after treatment prolong the treatment period. The aim of this prospective, randomized study was to compare the results of the widely used Limberg and Karydakis flap operations in recent years. The parameters that will be used in the comparison will be an infection, recurrence and wound decomposition.

ELIGIBILITY:
Inclusion Criteria:

* Pilonidal sinus disease

Exclusion Criteria:

* Other disease than pilonidal sinus disease.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-05-22 (Actual); Primary Completion 2021-05-22 (Estimated); Study Completion 2021-05-22 (Estimated)

PRIMARY OUTCOMES:
Postoperative recurrence | 1 month
  pain, swelling and redness in examination

SECONDARY OUTCOMES:
Postoperative infection | 1 week
  purulent drainage
Postoperative wound dehiscence | 1 week
  wound separation

CONTACTS AND LOCATIONS:
Overall Officials: ahmet gökhan güler, Principal Investigator — kahramanmarasSUI
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Onikisubat, Turkey (Türkiye)